CLINICAL TRIAL: NCT05924867
Title: Application of Plasma Activated Saline in Wound Treatment
Brief Title: Plasma Activated Saline in Wound Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-2021ZD03
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Wound; Wound Infection; Wound Heal
MeSH Terms: conditions — Wounds and Injuries; Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The wounds of participants in the postoperative incision infection group and ulcer infection group will be given plasma activated saline irrigation (100 ml plasma activated saline for every 10 cm2 wound), drainage, and wet compress. The wounds of participants in the fat liquefaction group will be uniformly rinsed with plasma saline for 5-10 min to clean the incision, then drained and suction with negative pressure.
  The researchers will determine the dressing change time according to the size of the patient's wound and the number of secretions, starting every day or every other day, and waiting for the incision to be fresh or less secretions at an interval of 2-3 days.
  Interventions: Other: plasma activated saline
- Control group (Active Comparator): The wounds of participants in the postoperative incision infection group and ulcer infection group will receive routine dressing change treatment, namely cleaning with chlorhexidine disinfectant (100 ml chlorhexidine disinfectant for every 10 cm2 wound area), drainage, bandaging. The wounds of participants in the fat liquefaction group will be receive conventional treatment, namely negative pressure sputum aspiration.
  The researchers will determine the dressing change time according to the size of the patient's wound and the number of secretions, starting every day or every other day, and waiting for the incision to be fresh or less secretions at an interval of 2-3 days.
  Interventions: Other: Routine nursing

INTERVENTIONS:
Other: plasma activated saline — The plasma activated normal saline used in the intervention was prepared by a self-made machine, and the safety of the plasma activated water produced by the machine has passed the national quality inspection.
  Arms: Intervention group
Other: Routine nursing — For postoperative incision infection group and infected ulcer group, conventional dressing change treatment was given, namely chlorhexidine disinfectant washing, drainage and bandaging; For the fat liquefaction group, conventional treatment was given, namely negative pressure suction.
  Arms: Control group

SUMMARY:
This is a prospective, open-label, randomized, parallel controlled clinical trial. The purpose of this study is to understand the application value of plasma-activated normal saline in the treatment of different types of wounds. The main questions it aims to answer are:

1. What is the effect of plasma activated normal saline in promoting wound healing of different types?
2. What is the safety of plasma activated normal saline in the treatment of wound surface? Subjects will be randomly divided into the intervention group and the control group. The intervention group will receive wound treatment with plasma activated normal saline, and the control group will receive routine dressing change treatment.

DETAILED DESCRIPTION:
As the population ages and antibiotic resistance increases, the chance of co-infection of various types of wounds increases greatly, resulting in prolonged wounds healing and eventually leading to bloodstream infections caused by germs, which can develop into life-threatening sepsis in severe cases. Plasma active saline is rich in reactive oxygen groups (ROS) and reactive nitrogen groups (RNS). It has good anti-inflammatory effect and is a potential new material to control wound infection and promote wound healing. Therefore, the purpose of this study was to apply plasma-activated water to different types of wounds and evaluate the effect of plasma-activated water on promoting healing of different types of wounds. And security issues in the application process.

This study is a prospective, open label, randomized, parallel controlled trial. This study is expected to include 162 subjects, including 46 patients with postoperative incision infection, 34 patients with postoperative incision fat liquefaction, and 82 patients with cutaneous infectious ulcer. The participants will be randomly divided into intervention group and control group by grouping randomized method. The intervention group will be treated with plasma activated water flushing and wet compress, and the control group will be treated with routine dressing change. The investigators will collect participants' wound conditions, blood, microbiological tests and other relevant indicators during treatment and follow-up.

To analyze the efficacy and safety of plasma-activated saline in the treatment of different wounds, the investigators will use independent sample T-test and K-M methods to compare the efficacy of the two groups, use descriptive analysis to represent the type and frequency of adverse events.

ELIGIBILITY:
1. Inclusion Criteria

   1. Group of postoperative incision infection

      * Age ≥18 years old, ≤75 years old, gender unlimited.
      * Clinical diagnosis of postoperative incision infection.
      * Must be no significant risk of head trauma or closed injury to the chest and abdomen.
      * Fully understand the study content and subjects' rights and interests, and sign the informed consent.
   2. Group of postoperative incision fat liquefaction

      * Age ≥18 years old, ≤75 years old, gender unlimited.
      * Clinical diagnosis of postoperative incision fat liquefaction.
      * Must be no incision infection or organ infection was involved in deep surgery, and no other serious complications occurred.
      * Must be no significant risk of head trauma or closed injury to the chest and abdomen.
      * Fully understand the study content and subjects' rights and interests, and sign the informed consent.
   3. Group of infectious ulcers

      * Age ≥18 years old, ≤75 years old, gender unlimited.
      * Clinical diagnosis of superficial skin ulcer infection caused by various causes, which can have one or more wounds.
      * The formation time of the wound surface exceeds 1 month.
      * Fully understand the study content and subjects' rights and interests, and sign the informed consent.
2. Exclusion Criteria

   * Allergic to multiple drugs, dressings, gels or materials used in this study.
   * Functional injury of cardiopulmonary system, with obvious risk of craniocerebral trauma or severe closed injury of chest and abdomen.
   * Severe malnutrition, hypoproteinemia, moderate to severe anemia.
   * Pregnant or lactating women (lactating female subjects can still be included if they agree to stop breastfeeding during the treatment period and within one week after the last medication).
   * Patients with active wound bleeding, poor mental condition and critical condition.
   * Poor glycemic control of diabetes mellitus; Severe malnutrition, hypoproteinemia, moderate and severe anemia.
   * The presence of inflammatory skin diseases, such as atopic dermatitis or eczema, that affect efficacy and safety evaluation.
   * Poor glycemic control of diabetes mellitus; Severe malnutrition, severe cardiopulmonary disease, hypertension, widespread local necrosis requiring immediate toe amputation.
   * Combined with anaerobic bacteria infection, wet gangrene, abdominal infection, hematogenous infection, and intra-articular infection.
   * Ulcers caused by diabetic feet and malignant tumors.
   * History of glucocorticoid use and anticoagulant drug use within 12 months before enrollment.
   * History of immune disease or immunosuppressant use.
   * Poor compliance due to cognitive impairment or mental illness.
   * Any conditions that the investigator considered might increase the risk to the subject or affect the evaluation of efficacy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
The trends in wound healing rate | 1 day up to 21 days
  Wound healing rate=Number of healing cases/total cases ×100%

SECONDARY OUTCOMES:
The number of participants with wound effusion | The indicators will be collected at day 1, 7, 14 and 21 after the start of treatment
  Observe whether there is fluid, pus and other exudation on the wound and the number of days when the effusion disappeared will be recorded.
The number of participants who tested positive for the etiology of wound exudates or extracts | The indicators will be collected at day 1, 7, 14 and 21 after the start of treatment.
  Check whether there is bacterial infection and infected strains on the wound.
Wound pain score | The indicators will be collected at day 1, 7, 14 and 21 after the start of treatment.
  Wound pain will be measured on the Visual Analogue Scale with a minimum score of 0 and a maximum score of 10 on the VAS, 0 indicating no pain at all, 10 indicating severe pain that is unbearable, and a higher score indicating more severe pain.
The number of adverse event | These indicators will be collected at 1, 7, 14, and 21 days after starting treatment, and at 1 week and 1 month after ending treatment.
  In this trial, any adverse medical event occurring within 30 days after the subject's signing of the informed consent to the final dose, regardless of whether there is a causal relationship with the test drug, is considered to be an adverse event. Adverse events and descriptions of all associated symptoms, such as time of occurrence, severity, duration, action taken, final outcome and outcome, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Chang, PhD, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirhaj M, Labbaf S, Tavakoli M, Seifalian A. An Overview on the Recent Advances in the Treatment of Infected Wounds: Antibacterial Wound Dressings. Macromol Biosci. 2022 Jul;22(7):e2200014. doi: 10.1002/mabi.202200014. Epub 2022 Apr 28. PMID 35421269
- [Background] Cheng B, Jiang Y, Fu X, Hao D, Liu H, Liu Y, Huang Z, Tan Q, Wang L, Hu D, Yang Y, Han C, Cheng Z, Ran X, Li Y. Epidemiological characteristics and clinical analyses of chronic cutaneous wounds of inpatients in China: Prevention and control. Wound Repair Regen. 2020 Sep;28(5):623-630. doi: 10.1111/wrr.12825. Epub 2020 Jun 25. PMID 32585756
- [Background] Kadam S, Shai S, Shahane A, Kaushik KS. Recent Advances in Non-Conventional Antimicrobial Approaches for Chronic Wound Biofilms: Have We Found the 'Chink in the Armor'? Biomedicines. 2019 Apr 30;7(2):35. doi: 10.3390/biomedicines7020035. PMID 31052335
- [Background] Sen CK. Human Wound and Its Burden: Updated 2020 Compendium of Estimates. Adv Wound Care (New Rochelle). 2021 May;10(5):281-292. doi: 10.1089/wound.2021.0026. PMID 33733885
- [Background] Bernhardt T, Semmler ML, Schafer M, Bekeschus S, Emmert S, Boeckmann L. Plasma Medicine: Applications of Cold Atmospheric Pressure Plasma in Dermatology. Oxid Med Cell Longev. 2019 Sep 3;2019:3873928. doi: 10.1155/2019/3873928. eCollection 2019. PMID 31565150
- [Background] Brany D, Dvorska D, Halasova E, Skovierova H. Cold Atmospheric Plasma: A Powerful Tool for Modern Medicine. Int J Mol Sci. 2020 Apr 22;21(8):2932. doi: 10.3390/ijms21082932. PMID 32331263
- [Background] Smolkova B, Frtus A, Uzhytchak M, Lunova M, Kubinova S, Dejneka A, Lunov O. Critical Analysis of Non-Thermal Plasma-Driven Modulation of Immune Cells from Clinical Perspective. Int J Mol Sci. 2020 Aug 28;21(17):6226. doi: 10.3390/ijms21176226. PMID 32872159
- [Background] Rezaei F, Vanraes P, Nikiforov A, Morent R, De Geyter N. Applications of Plasma-Liquid Systems: A Review. Materials (Basel). 2019 Aug 27;12(17):2751. doi: 10.3390/ma12172751. PMID 31461960
- [Background] Zhai S, Xu M, Li Q, Guo K, Chen H, Kong MG, Xia Y. Successful Treatment of Vitiligo with Cold Atmospheric Plasma-Activated Hydrogel. J Invest Dermatol. 2021 Nov;141(11):2710-2719.e6. doi: 10.1016/j.jid.2021.04.019. Epub 2021 May 21. PMID 34029575
- [Background] Tanaka H, Bekeschus S, Yan D, Hori M, Keidar M, Laroussi M. Plasma-Treated Solutions (PTS) in Cancer Therapy. Cancers (Basel). 2021 Apr 6;13(7):1737. doi: 10.3390/cancers13071737. PMID 33917469
- [Background] Lee HR, Kang SU, Kim HJ, Ji EJ, Yun JH, Kim S, Jang JY, Shin YS, Kim CH. Liquid plasma as a treatment for cutaneous wound healing through regulation of redox metabolism. Cell Death Dis. 2023 Feb 13;14(2):119. doi: 10.1038/s41419-023-05610-9. PMID 36781835
- [Background] Xu D, Wang S, Li B, Qi M, Feng R, Li Q, Zhang H, Chen H, Kong MG. Effects of Plasma-Activated Water on Skin Wound Healing in Mice. Microorganisms. 2020 Jul 21;8(7):1091. doi: 10.3390/microorganisms8071091. PMID 32708347
- [Background] Kim S, Kim CH. Applications of Plasma-Activated Liquid in the Medical Field. Biomedicines. 2021 Nov 16;9(11):1700. doi: 10.3390/biomedicines9111700. PMID 34829929
- [Background] Jang Y, Bok J, Ahn DK, Kim CK, Kang JS. Human Trial for the Effect of Plasma-Activated Water Spray on Vaginal Cleaning in Patients with Bacterial Vaginosis. Med Sci (Basel). 2022 Jun 18;10(2):33. doi: 10.3390/medsci10020033. PMID 35736353
- [Result] Liu Z, Dumville JC, Norman G, Westby MJ, Blazeby J, McFarlane E, Welton NJ, O'Connor L, Cawthorne J, George RP, Crosbie EJ, Rithalia AD, Cheng HY. Intraoperative interventions for preventing surgical site infection: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2018 Feb 6;2(2):CD012653. doi: 10.1002/14651858.CD012653.pub2. PMID 29406579
- [Result] Leren L, Johansen EA, Eide H, Sorum Falk R, Ljosa TM. Prevalence and factors associated with ulcer-related pain in persons with chronic leg ulcers-an explorative study. J Clin Nurs. 2021 Sep;30(17-18):2732-2741. doi: 10.1111/jocn.15787. Epub 2021 May 5. PMID 33951254
- [Result] Liu HR, Yang P, Han S, Zhang Y, Zhu HY. The application of enhanced recovery after surgery and negative-pressure wound therapy in the perioperative period of elderly patients with colorectal cancer. BMC Surg. 2021 Sep 6;21(1):336. doi: 10.1186/s12893-021-01331-y. PMID 34488699
- [Result] Zhang J, Qu K, Zhang X, Wang B, Wang W, Bi J, Zhang S, Li Z, Kong MG, Liu D, Liu C. Discharge Plasma-Activated Saline Protects Against Abdominal Sepsis by Promoting Bacterial Clearance. Shock. 2019 Jul;52(1):92-101. doi: 10.1097/SHK.0000000000001232. PMID 30028781
- [Result] Seidel D, Diedrich S, Herrle F, Thielemann H, Marusch F, Schirren R, Talaulicar R, Gehrig T, Lehwald-Tywuschik N, Glanemann M, Bunse J, Huttemann M, Braumann C, Heizmann O, Miserez M, Kronert T, Gretschel S, Lefering R. Negative Pressure Wound Therapy vs Conventional Wound Treatment in Subcutaneous Abdominal Wound Healing Impairment: The SAWHI Randomized Clinical Trial. JAMA Surg. 2020 Jun 1;155(6):469-478. doi: 10.1001/jamasurg.2020.0414. PMID 32293657